CLINICAL TRIAL: NCT03180866
Title: Evaluation of Efficacy, Duration of Remission and Safety of a Light and Occlusive Patch Therapy for Plaque Psoriasis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Illumicure Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: L-003
Record Dates: First submitted 2017-05-09; First posted 2017-06-08 (Actual); Last update posted 2017-06-08 (Actual); Status verified 2017-06

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: The subject will act as their own control as one target plaque will receive treatment and one will not. This information will not be made available to the Investigators or the bio-statistician.
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Non-treatment Control (No Intervention): Control arm will not have any intervention
- Luma Light System (Experimental): The experimental arm will be a combination of an occlusive dressing and NBUVB light.
  Interventions: Device: Luma Light System

INTERVENTIONS:
Device: Luma Light System — The Luma Light System combines a NBUVB light with an occlusive dressing.
  Arms: Luma Light System

SUMMARY:
This is a proof of concept, investigator blinded study to evaluate the efficacy and safety of a novel combination of a home narrow band ultraviolet B (NBUVB) lamp with an occlusive dressing in adult subjects with mild to moderate psoriasis vulgaris. Two interpatient arms will be used to compare the efficacy of combination of NBUVB with an occlusive dressing (active) to no treatment (control). 32 patients will be enrolled in this 30 week study.

DETAILED DESCRIPTION:
This is a multi-center, investigator blinded, randomized study designed to assess the efficacy, duration of effect, safety and tolerability of Luma Light System for plaque psoriasis. Two selected areas to be treated will be determined by the Investigator at Baseline. Excluded areas include the palms, the soles of the feet, the intertriginous areas, the knee, the elbow, the face and the scalp. Target Plaque Assessment (TPA), tolerability assessment and any adverse events (AEs) will be obtained at each visit. The subject may use topical prescriptions (steroids, vitamin D analogs, retinoids, etc.) for non-target plaques during this trial with approval of the investigator as long as they keep a 1" border around the target plaques where no prescription topical is applied. Any treatment that is not part of the trial that the subject uses for psoriasis should be noted in the subject's file.

Start of Observation Phase with Screening Visit: Subjects will be given an IRB approved consent to read and sign at the screening Visit. No study related procedures will be performed prior to signing this consent. The Investigator will review the inclusion/exclusion criteria, evaluate the Subject's medical history, before determining the Subject's eligibility to participate in the study. A pregnancy test will be performed for all females of childbearing potential at the Screening Visit. Prior to the trial start, each subject will undergo a minimum 2 weeks or maximum of 13 weeks Observation Phase (starting with Visit 1 Screening) during which the subject will be supplied a standard cleanser and lotion in order to evaluate the stability of the plaque severity prior to entering the Active Treatment Phase. The Observation Phase will be up to 13 weeks if the subject needs to taper off an oral medication or biologic (see Washout and Excluded Medications section).

Start of Active Treatment Phase with Baseline Visit: If the Subject is determined to be eligible for the study, he/she will return to the clinic for the Baseline Visit. At this visit inclusion/exclusion criteria will be confirmed, patient will be enrolled in the study, randomization of the plaques will occur and baseline assessments will be performed including TPA. The test product will be dispensed, the user will be trained on how to use the product and the first treatment will be applied.

The Active Treatment Phase will be 6 weeks or until target plaque has cleared, whichever comes first. During the Active Treatment Phase, the plaque randomized to Arm B will receive the active occlusive hydrogel patch and will be changed every 5 days or less as needed. During the Active Treatment Phase, the plaque randomized to Arm A will receive the window patch and replaced as needed. The light will be applied to the target plaque assigned to Arm B every day with the hydrogel patch in place. The subject will return to the clinic every two weeks (Visit 3, 4 and 5) for assessments. Subjects who terminate early will be asked to complete all Week 6/ET assessments prior to commencement of any alternative therapy for psoriasis (if possible). Subjects who discontinue from the study during the Active Treatment Phase may be replaced and only will be followed if an AE is present.

Start of Follow-up Phase: Subjects will return for efficacy and safety follow-up visits at 8 week intervals after the Active Treatment Phase for 24 weeks (Visit 6, 7 and 8) to assess durability of remission. If subject decides to start active treatment with a prescription product on a plaque that was treated during the Active Treatment Phase (not including supplied lotion and cleanser, shampoos for hair or their normal topical therapeutic products to psoriatic areas that are not part of the study treatment areas) then that target plaque will no longer considered to be in remission. No systemic treatments will be allowed during the Follow-up Phase but if the subject or physician determines that it is necessary, the subject will no longer be considered in remission at the time of commencement of the systemic treatment. If the subject uses a prescription product on a target plaque or starts a systemic treatment, the investigator will capture why this occurs.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female of any race, greater than 18 years of age.
2. Verbal and written informed consent obtained from the subject.
3. Has a clinical diagnosis of plaque psoriasis at the Screening and Baseline visits.
4. Has an IGA score of 2 to 4 that is consistent between the Screening and Baseline visits.
5. TPA score of 5-12 and a score of at least 1 for each of the 3 different psoriasis signs and symptoms (erythema, plaque elevation, and scaling) at the baseline visits.
6. Has at least 2 plaques of at least 6cm by 3cm with TPA scores not differing from each other by a score of more than 1 that are at least 2 inches apart at the baseline visit.
7. Is in good general health as determined by the Investigator based on the subject's medical history.
8. Females of childbearing potential must have negative urine or blood pregnancy test results. Females of childbearing potential agree to use acceptable methods of contraception from the screening visit continuously until 30 days after end of treatment.
9. Subject agrees to use only the Sponsor provided cleanser and lotion during the study phase unless given permission by Investigator to use other topicals on non-target plaques.
10. Subject is willing and able to return for all study visits.

Exclusion Criteria:

1. Presence of psoriasis that was previously treated with prescription medications prior to the Screening visit and was non-responsive to treatment, as determined by the Investigator.
2. Presence of any concurrent skin condition that could interfere with the evaluation of the study device, as determined by the Investigator.
3. Female who is pregnant, nursing an infant, or planning a pregnancy during the Active Treatment Phase.
4. Treatment with any investigational drug or device within 2 weeks or 5 half-lives (whichever is longer) prior to the Baseline visit, or concurrent participation in another clinical trial with an investigational drug or device.
5. History of melanoma.
6. Subject has any medical, social or psychological conditions that, in the opinion of the Investigator, preclude them from receiving the pre-treatment, required treatment, and post-treatment procedures and evaluations.
7. Subject has known allergy or adverse reaction to skin adhesives or hydrogels or coal tar.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2016-12; Primary Completion 2018-03 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
Target Plaque Assessment (TPA) at 6 weeks | 6 weeks
  Local efficacy will be evaluated with a 0-4 point scale for three signs and symptoms of psoriasis: erythema, plaque elevation, and scaling. Change in TPA score will be used to measure the efficacy of the Luma Light System at 6 weeks after treatment initiation compared to control. TPA change scores will be computed by subtracting scores at baseline from scores at 6 weeks. It is hypothesized that the decline in TPA scores will be greater for the Luma Light System (Arm B) than for the control (Arm A).

SECONDARY OUTCOMES:
Frequency and severity of device and / or procedure related adverse events | 6 weeks
  Profile the safety of the Luma Light System (Arm B) in terms of the frequency and severity of device and / or procedure related adverse events. Evaluation of adverse events, including significant changes from baseline in cutaneous tolerability (burning/stinging, pain, and pruritus) of a combination of a home NBUVB lamp with an occlusive hydrogel patch (Arm B).
TPA at 2, 4, 22 and 30 weeks | 2, 4, 22 and 30 weeks
  TPA measurement of efficacy at weeks 2, 4, 14, 22 and 30 of Luma Light System (Arm B) compared to control (Arm A). TPA change scores will be computed by subtracting scores at baseline from scores at each specified study visit.
Duration of remission | 30 weeks
  Duration of remission of plaques of the Luma Light System (Arm B) compared to control (Arm A). Duration of remission is defined by days between plaque clearing and whichever comes first: either the 30 week visit 8, withdrawal from the study for any reason or follow-up TPA score of 2 or higher. A plaque is considered cleared with a scale and thickness score of 0 and an erythema score of 1 or 0. If a plaque does not reach this score the remission duration will be zero.
Subject Satisfaction | 4 weeks
  Subject satisfaction with treatment and perceived plaque improvement of the Luma Light System (Arm B) at 4 weeks compared to control (Arm A).
Compliance | 6 weeks
  Compliance to Luma Light System (Arm B) in terms of percent daily treatments delivered.
TPA less than 2 at 4 weeks | 4 weeks
  Percentage of subjects who reach a TPA score of less than 2 in treatment Arms A and B in 4 and 6 weeks.
TPA less than 2 at 6 weeks | 6 weeks
  Percentage of subjects who reach a TPA score of less than 2 in treatment Arms A and B
Subject Satisfaction | 6 weeks
  Subject satisfaction with treatment and perceived plaque improvement of the Luma Light System (Arm B) at 6 weeks compared to control (Arm A).

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Redwood Dermatology Research, Santa Rosa, California
  - Dermatology Associates of Knoxville, PC, Knoxville, Tennessee
  - Texas Dermatology and Laser Specialists, San Antonio, Texas
  - Jordan Valley Dermatology Center, West Jordan, Utah

IPD SHARING:
Plan to Share IPD: No